CLINICAL TRIAL: NCT00227565
Title: Phase II Trial of Pemetrexed Disodium and Carboplatin in Previously Untreated Extensive Stage Small Cell Lung Cancer
Brief Title: Pemetrexed Disodium and Carboplatin in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0423; NCI-2012-02671 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000442866 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Pemetrexed; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pemetrexed + carboplatin + radiation (Experimental): Patients receive pemetrexed disodium IV over 10 minutes and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who develop progressive disease in the CNS only may receive whole-brain radiotherapy and then continue chemotherapy after completion of whole-brain radiotherapy for up to 6 courses.
  After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 4 years.
  Interventions: Drug: carboplatin; Drug: pemetrexed disodium; Radiation: radiation

INTERVENTIONS:
Drug: carboplatin
Drug: pemetrexed disodium
Radiation: radiation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving pemetrexed disodium together with carboplatin works in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete and partial response rates in patients with previously untreated, extensive-stage small cell lung cancer treated with pemetrexed disodium and carboplatin.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine, preliminarily, the survival of patients treated with this regimen.
* Determine, preliminarily, the response rate in patients 70 years and older treated with this regimen.
* Determine, preliminarily, the toxicity of this regimen in patients 70 years and older.

OUTLINE: This is a multicenter study. Patients are stratified according to age (< 70 years vs ≥ 70 years).

Patients receive pemetrexed disodium IV over 10 minutes and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who develop progressive disease in the CNS only may receive whole-brain radiotherapy and then continue chemotherapy after completion of whole-brain radiotherapy for up to 6 courses.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 4 years.

PROJECTED ACCRUAL: Approximately 77 patients at least 46 who are < 70 years of age and at least 24 who are ≥ 70 years of age) will be accrued for this study within 20-26 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer

  * Previously untreated disease
  * No mixed histology
* Extensive-stage disease

  * Clinically significant effusions (e.g., symptomatic pleural effusion) must be drained prior to treatment
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No symptomatic, untreated, or uncontrolled CNS metastases

  * CNS metastases previously treated with whole-brain radiotherapy allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) OR
* Direct bilirubin normal
* ALT and AST ≤ 3 times ULN (5 times ULN if there is liver involvement)

Renal

* Creatinine clearance ≥ 45 mL/min

Cardiovascular

* No angina pectoris
* No congestive heart failure within the past 3 months, unless ejection fraction > 40%
* No cardiac arrhythmia
* No myocardial infarction within the past 3 months
* No hypertension, including labile hypertension

Pulmonary

* No interstitial pneumonia
* No extensive and symptomatic interstitial fibrosis of the lung

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of poor compliance with antihypertensive medication
* Able to take folic acid, cyanocobalamin (vitamin B_12) supplementation, or dexamethasone
* No uncontrolled diabetes
* No serious condition that would preclude study participation
* No clinically significant infection
* No significant traumatic injury
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer

  * Low-grade (Gleason score ≤ 6), localized prostate cancer allowed even if diagnosed < 5 years prior to study entry
* No seizure disorder
* No other severe and/or uncontrolled medical condition

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy
* No concurrent immunomodulating agents

Chemotherapy

* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* See Disease Characteristics
* Prior palliative radiotherapy allowed

  * No prior palliative radiotherapy to the chest except for ≤ 3 fractions for superior vena cava syndrome
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery* (i.e., laparotomy) or open biopsy
* More than 2 weeks since prior minor surgery* NOTE: *Insertion of a vascular access device is not considered major or minor surgery

Other

* More than 4 weeks since prior investigational therapy
* No concurrent Hypericum perforatum (St. John's wort)
* No concurrent inducers or inhibitors of CYP3A4
* No concurrent medications that are metabolized by CYP3A4
* No aspirin dose ≥ 1.3 grams per day for ≥ 10 days prior to and after study treatment
* No other concurrent cytostatic or cytotoxic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Proportion of confirmed-tumor response | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: James R. Jett, MD, Study Chair — Mayo Clinic
Locations (148):
- United States (148):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Albert Lea Cancer Center at Albert Lea Medical Center, Albert Lea, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Result] Chee CE, Jett JR, Bernath AM Jr, Foster NR, Nelson GD, Molina J, Nikcevich DA, Steen PD, Flynn PJ, Rowland KM Jr. Phase 2 trial of pemetrexed disodium and carboplatin in previously untreated extensive-stage small cell lung cancer, N0423. Cancer. 2010 May 15;116(10):2382-9. doi: 10.1002/cncr.24967. PMID 20209614
- [Result] Jett JR, Bernath AM, Foster NR, et al.: Phase II trial of pemetrexed (P) and carboplatin (C) in previously untreated extensive stage disease small cell lung cancer (ED-SCLC): A NCCTG Study. [Abstract] J Clin Oncol 26 (Suppl 15): A-8066, 2008.